CLINICAL TRIAL: NCT04912843
Title: A Phase 1/2/3, Multi-center, Two-part Clinical Trial to Evaluate the Safety and Efficacy of Gene Therapy for Leber's Hereditary Optic Neuropathy (LHON) Associated With ND4 Mutation
Brief Title: Gene Therapy Clinical Trial for the Treatment Of Leber's HereDitary Optic Neuropathy
Acronym: GOLD
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Wuhan Neurophth Biotechnology Limited Company (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NFS-01-101
Record Dates: First submitted 2021-05-13; First posted 2021-06-03 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Leber's Hereditary Optic Neuropathy (LHON)
MeSH Terms: conditions — Optic Atrophy, Hereditary, Leber

STUDY DESIGN:
Intervention Model Description: Part 1: Dose-Finding At the dose-finding part, the principle is that the Safety Review Committee (SRC) will determine whether to make dose adjustment based on the safety data of the starting dose in Part 1. The recommended dose (safe and effective dose) of the Part 2 study will be determined jointly by the SRC, IDMC, sponsor and the drug regulatory authority after the interim analysis in Part 1 is completed.
  Part 2 :
  First Stage: safety run-in phase:
  The safety run-in phase of Part 2 will enroll 6 evaluable subjects (including at least 1 minor subject aged ≥ 12 years and < 18 years) aged ≥ 12 years and ≤ 75 years at the dose determined in Part 1, namely 4.5 x 109 vg, 0.05 mL eye/dose (high dose) and monitor the safety for at least 6 weeks. If there is no new safety concern evaluated by the SRC, the randomized, double-blind, sham-injection control study can be initiated.
  Second Stage: randomized, double-blind, sham-injection control study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 1: Dose-Finding: open label；12 subjects Part 2: First Stage: safety run-in phase: open label；6 subjects Part 2: Second Stage: randomized, double-blind, sham-injection; 90 subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NR082 injection (Experimental): 0.5E9 viral genomes (vg), 0.05 mL eye/dose ,single-dose,only one eye per subject; 1.5E9 viral genomes (vg), 0.05 mL eye/dose single-dose,only one eye per subject; 4.5E9 viral genomes (vg) , 0.05 mL eye/dose single-dose,only one eye per subject Part 1: Dose-Finding；The recommended dose (safe and effective dose) of the Part 2 study will be determined jointly by the SRC, IDMC, sponsor and the drug regulatory authority after the interim analysis in Part 1 is completed.
  Interventions: Drug: NR082 injection
- sham-injection (Sham Comparator): Part2.Second Stage: randomized, double-blind, sham-injection control study One eye of each participant will undergo sham injection. Sham intravitreal injection will be performed by applying pressure to the eye at the location of a typical intravitreal injection procedure using the blunt end of a syringe without a needle.
  Interventions: Device: Sham Injection

INTERVENTIONS:
Drug: NR082 injection — Intravitreal injection（IVT）
  Arms: NR082 injection
Device: Sham Injection — Sham Intravitreal Injection
  Arms: sham-injection

SUMMARY:
The objective of this clinical study is to select the optimal dose and evaluate the safety and efficacy of NR082 in treatment of LHON caused by mitochondrial ND4 gene mutation. Part 1 (Phase 1/2) is a safety dose-finding study, which will enroll subjects aged ≥ 18 years old and ≤ 75 years old to receive a single unilateral intravitreal (IVT) injection of NR082 to observe its safety and efficacy. In Part 2 (Phase 3) of the clinical study, the dose recommended after the end of Part 1 is used to further verify the safety and efficacy of the study drug. Part 2 of the study is divided into the safety run-in phase and the randomized, double-blind and control study. Subjects aged ≥ 12 years and ≤ 75 years will be enrolled in the Part 2. The run-in phase will enroll 6 evaluable subjects. After monitoring for at least 6 weeks, if no new safety signals are observed, the clinical trial will enter the randomized, double-blind and control study phase upon approval by the Safety Review Committee(SRC). The clinical manifestation of all subjects is reduced visual acuity caused by LHON associated with ND4 mutation, and central laboratory test showed G11778A mutation (a CLIA-certified laboratory), while the reduced visual acuity lasted for > 6 months and < 10 years.

DETAILED DESCRIPTION:
Part 1: Dose-Finding At the dose-finding part, the principle is that the Safety Review Committee (SRC) will determine whether to make dose adjustment based on the safety data of the starting dose in Part 1. The recommended dose (safe and effective dose) of the Part 2 study will be determined jointly by the SRC, IDMC, sponsor and the drug regulatory authority after the interim analysis in Part 1 is completed.

The starting dose in Part 1 is 1.5 × 109 vg, 0.05 mL eye/dose. The safety of the starting dose will be reviewed by the SRC and the dose escalation or de-escalation will be recommended by the SRC.

The safety of the starting dose will first be performed in 6 evaluable subjects.

Part 2 (including the safety run-in phase and the randomized, double-blind and sham-injection control study):

First Stage: safety run-in phase:

The safety run-in phase of Part 2 will enroll 6 evaluable subjects (including at least 1 minor subject aged ≥ 12 years and < 18 years) aged ≥ 12 years and ≤ 75 years at the dose determined in Part 1, namely 4.5 x 109 vg, 0.05 mL eye/dose (high dose) and monitor the safety for at least 6 weeks. If there is no new safety concern evaluated by the SRC, the randomized, double-blind, sham-injection control study can be initiated.

Second Stage: randomized, double-blind, sham-injection control study:

The randomized, double-blind, sham-injection control study of Part 2 is to verify the efficacy and safety of NR082 in LHON caused by mitochondrial gene ND4 mutation at the dose determined in Part 1 of the study, namely 4.5 x 109 vg, 0.05 mL eye/dose (high dose). This part is divided into the NR082 treatment group and the control group (sham-injection group).

ELIGIBILITY:
Inclusion Criteria Age

1. Age at signing of informed consent form

   1. In Part 1, the age of the subjects must be ≥ 18 years old and ≤ 75 years old
   2. In Part 2, the age of the subjects must be ≥ 12 years old and ≤ 75 years old, and the 6 evaluable subjects must be monitored for at least 6 weeks during the safety run-in phase. If SRC believes that there is no safety issue, the randomized double-blind control study will be initiated Subject Type and Disease Characteristics
2. The clinical manifestation caused by LHON is vision loss, with a visual acuity of ≥ 0.5 LogMAR in BCVA in either eye
3. The genotype test result is that there is G11778A mutation in ND4 gene, and there are no other primary LHON-associated mutations in the mitochondrial DNA (mtDNA) (ND1[G3460A] or ND6[T14484C]) (confirmed by a CLIA-certified international laboratory)
4. The duration of vision loss in the eye with worse visual acuity lasted > 6 months and < 10 years at screening
5. Pupils can be adequately dilated for a comprehensive eye examination and visual acuity test
6. Each eye of the subject must maintain the VA determined by manual visual acuity test (≤ 2.3 LogMAR) as defined in the ocular/vision examination manual (operating manual for optometry and VA examinations) in this study
7. Sign the written informed consent form and willing to comply with the clinical study protocol Sex
8. Male or female

   1. Male subjects:

      • A male subject must agree to take contraceptive measures at least 6 months after the treatment visit, see Appendix 5 for details
   2. Female subjects:

      * A female subject is eligible to participate if she is not pregnant (see Appendix 5), not breastfeeding, and at least one of the following conditions applies:

   i) Not a woman of childbearing potential (WOCBP) as defined in Appendix 5 or ii) A WOCBP who agrees to follow the contraception guidance in Appendix 5 for at least 6 months after the treatment visit Informed Consent
9. Written informed consent form must be obtained from the subject or his/her parent/legal guardian (if the subject is under 18 years of age) (Part 2) before any study-related procedures are performed (see Section 10.2) If the subject is legally identified as blind (>1.0 LogMARor decimal acuity meter reading < 0.1), an impartial witness must be present throughout the informed consent process and discussion process.

Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from the study:

1. Any known allergy and/or hypersensitivity to the study drug or its constituents
2. Contraindication to IVT injection in any eye
3. IVT drug delivery to any eye within 30 days prior to the screening visit
4. History of vitrectomy in either eye
5. Narrow anterior chamber angle in any eye contra-indicating pupillary dilation
6. Presence of disorders or diseases of the eye or adnexa, excluding LHON, which may interfere with visual or ocular assessments, including spectral-domain optical coherence tomography (FD-OCT), during the study
7. Presence of known/documented mutations, other than the LHON-related mutation, which are known to cause pathology of the optic nerve, retina or afferent visual system
8. Presence of systemic or ocular/vision diseases, disorders or pathologies, other than LHON, known to cause or be associated with vision loss, or whose associated treatment(s) or therapy(ies) is/are known to cause or be associated with vision loss
9. Presence of optic neuropathy from any cause other than LHON
10. Presence of illness or disease that, in the opinion of the investigator, include symptoms and/or the associated treatments that can alter visual function, for instance cancers or pathology of the CNS, including multiple sclerosis (diagnosis of multiple sclerosis must be based on the 2010 Revisions to the McDonald Criteria) (Polman et al., 2011), and/or diseases or conditions that affect the safety of subjects participating in the study
11. History of recurrent uveitis (idiopathic or immune-related) or active ocular inflammation
12. Participated in another clinical study and receive IP within 90 days prior to the screening visit

    a) Exceptions: Subjects who have completed the clinical study of idebenone as IP within 90 days prior to the screening visit, and has completely discontinued idebenone at least 7 days prior to dosing are still eligible to participate in the study.
13. Any eye has previously received ocular gene therapy
14. Subjects who refused to stop using idebenone
15. Have undergone ocular surgery of clinical relevance (per investigator's assessment) within 90 days prior to the screening visit
16. Female subjects who are breastfeeding or plan to breastfeed within the first 6 months after the administration of NR082 Injection
17. History of drug or alcohol abuse (including heavy smoking, i.e. > 20 cigarettes per day or > 20 pack-years [equivalent to one pack a day for 20 years or 2 packs a day for 10 years])
18. Subjects with positive human immunodeficiency virus (HIV), syphilis and HCV antibodies are excluded; subjects who have clinically significant active infection requiring treatment as shown by hepatitis B test (defined as positive hepatitis B core antibody [HBcAb] or hepatitis B surface antigen [HBsAg], hepatitis B virus deoxyribonucleic acid (HBV-DNA) >1,000 copies /mL or >lower limit of quantitative detection with the local laboratory method) will be excluded
19. Unable to tolerate or unable or unwilling to comply with all the protocol requirements
20. Subjects from the study site fail to comply with or do not agree to comply with local and institutional guidelines for suspected 2019 novel coronavirus (COVID-19) infection/testing
21. Any other exclusions determined by the investigator

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2021-06-18 (Actual); Primary Completion 2024-02-29 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of NR082 at different doses | Part 1 (Phase1/2): 12 weeks
  Incidence rates of AEs, SAEs and DLTs within 12 weeks after injection of NR082 at different doses
Safety after NR082 treatment among subjects 12 ≤ aged ≤ 75 years | Part 2 (Stage 1) : 6 weeks
  Incidence rates of AEs and SAEs within 6 weeks after NR082 treatment
Efficacy of NR082 in study eye | Part 2 (Stage 2): 52 weeks
  Proportion of ≥ 0.3 LogMAR from baseline in BCVA in the study eye in the NR082 treatment and the sham-injection at Week 52 after treatment

SECONDARY OUTCOMES:
The efficacy and safety following intravitreal injection of NR082 at different doses | Part 1 (Phase1/2), Part 2 (Stage 1 and Stage 2): Week 2, 6, 12, 26, 40 and 52
  Improvent and mean change from baseline in BCVA; Change from baseline in visual field, contrast sensitivity and visual evoked potential
Further assess the efficacy and safety following intravitreal injection of NR082 at different doses | Part 1 (Phase1/2) and Part 2 (Stage 1): At Weeks 26, 40 and 52
  Descriptions of safety evaluation at Weeks 26, 40 and 52
Immunogenicity and vector shedding/biodistribution | Part 1 (Phase1/2), Part 2 (Stage 1 and Stage 2): Week 2, 6, 12, 26, 40 and 52
  Assessment of cell immunity, humoral immunity, vector DNA shedding in tears (both eyes) and biodistribution in whole blood
The change in quality of life from baseline | Part 1 (Phase1/2), Part 2 (Stage 1 and Stage 2): Week 2, 26 and 52
  Change from baseline in VFQ-25 and SF-36
Morphological improvement after NR082 treatment | Part 1 (Phase1/2), Part 2 (Stage 1 and Stage 2): Week 2, 6, 12, 26, 40 and 52
  Change from baseline in RNFL, GCL and IPL thickness in the study eye
Safety and efficacy of NR082 caused by mitochondrial gene ND4 mutation | Part 2 (Stage 2): Week 2, 6, 12, 26, 40 and 52
  Incidence rates of AEs and SAEs between the NR082 treatment group and the sham-injection group (ocular and non-ocular)

CONTACTS AND LOCATIONS:
Overall Officials: Bin Li, MD, Study Chair — Wuhan Neurophth Biotechnology Limited Company
Locations (1):
- Beijing Tongren Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No